CLINICAL TRIAL: NCT07243444
Title: Efficacy of Home-Based Telerehabilitation Versus Center-Based Cardiac Rehabilitation on Cardiopulmonary Function and Exercise Capacity in Patients After Coronary Artery Bypass Grafting: A Randomized Controlled Trial
Brief Title: Home-Based Versus Center-Based Cardiac Rehabilitation After CABG Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yan Liu, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S00775-1
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home-Based Telerehabilitation (HBTCR) Group (Experimental): Participants received a personalized 12-week cardiac rehabilitation program to perform at home. They were provided with a wearable heart rate monitor and used a mobile application to log their exercise sessions and vital signs. A rehabilitation team remotely monitored their progress and communicated weekly via phone or video call.
  Interventions: Behavioral: Structured Exercise Program
- Center-Based Cardiac Rehabilitation (CBCR) Group (Active Comparator): Participants attended supervised cardiac rehabilitation sessions at the hospital's rehabilitation center three times per week for 12 weeks. Each session included warm-up, aerobic exercise, resistance training, and cool-down under the direct supervision of a healthcare team.
  Interventions: Behavioral: Structured Exercise Program
- Control Group (Sham Comparator): Participants received usual care, which included routine follow-up appointments and standard health education delivered through verbal instructions and printed pamphlets. They did not participate in a structured or monitored exercise program.
  Interventions: Behavioral: Standard Health Education

INTERVENTIONS:
Behavioral: Structured Exercise Program — A 12-week comprehensive cardiac rehabilitation program. The exercise prescription (frequency, intensity, duration, type) was based on a baseline cardiopulmonary exercise test, typically starting at 40-60% of heart rate reserve and increasing progressively. The program included aerobic and resistance training components. This intervention was delivered either remotely (HBTCR group) or in-person (CBCR group), three times per week.
  Arms: Center-Based Cardiac Rehabilitation (CBCR) Group; Home-Based Telerehabilitation (HBTCR) Group
Behavioral: Standard Health Education — Participants received routine follow-up and standard health education pamphlets covering topics such as medication adherence, diet, and general advice on physical activity, without a structured or monitored exercise plan.
  Arms: Control Group

SUMMARY:
This randomized controlled trial was designed to compare the efficacy of a 12-week home-based telerehabilitation (HBTCR) program against traditional center-based cardiac rehabilitation (CBCR) and usual care in patients who have undergone coronary artery bypass grafting (CABG). The primary goal was to assess changes in cardiopulmonary function, measured by peak oxygen consumption (VO₂ peak), and exercise capacity, measured by the 6-minute walk test (6MWT), to determine if HBTCR is a viable alternative to CBCR.

DETAILED DESCRIPTION:
While cardiac rehabilitation (CR) is a Class IA recommendation for patients after coronary artery bypass grafting (CABG) to improve long-term outcomes, participation in traditional center-based programs (CBCR) is low due to barriers like travel, cost, and scheduling. Home-based telerehabilitation (HBTCR) emerges as a potential solution. This study was a three-arm, prospective, single-center randomized controlled trial to rigorously evaluate if a structured HBTCR program is as effective as CBCR. A total of 110 patients, 4-8 weeks post-CABG, were randomized into three groups: HBTCR, CBCR, or a control group receiving usual care with educational pamphlets. The HBTCR group performed prescribed exercises at home, using wearable monitors and a mobile app, with weekly remote monitoring by a rehabilitation team. The CBCR group attended supervised sessions at the hospital three times a week. The control group received standard follow-up and educational materials. The interventions lasted 12 weeks, with assessments of cardiopulmonary function, exercise capacity, cardiac function, psychological status, and quality of life conducted at baseline and at 12 weeks. The study aimed to provide robust evidence for HBTCR as an effective alternative model of care for post-CABG rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30 to 75 years.
* Had undergone Coronary Artery Bypass Grafting (CABG) 4 to 8 weeks prior.
* In a stable clinical condition.
* Able to provide written informed consent.
* No cognitive impairments.

Exclusion Criteria:

* Acute decompensated heart failure.
* Severe physical comorbidities (e.g., fractures, severe hearing impairment) that would preclude participation in an exercise program.
* Recent stroke or pulmonary embolism.
* Significant hepatic or renal dysfunction.
* Unstable angina.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Peak Oxygen Consumption (VO₂ peak) | Baseline, 12 weeks
  Measured in mL/kg/min by cardiopulmonary exercise testing (CPET) on a treadmill using a symptom-limited protocol. The change from baseline to 12 weeks was assessed.
Change in 6-Minute Walk Distance (6MWD) | Baseline, 12 weeks
  Measured in meters, assessing the maximum distance a patient can walk in 6 minutes on a flat, hard surface. The change from baseline to 12 weeks was assessed.

SECONDARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) | Baseline, 12 weeks
  Assessed as a percentage (%) by transthoracic echocardiography.
Change in Forced Expiratory Volume in 1 second to Forced Vital Capacity Ratio (FEV1/FVC) | Baseline, 12 weeks
  Measured by spirometry to assess pulmonary function.
Change in Psychological Status (Anxiety) | Baseline, 12 weeks
  Assessed using the Hamilton Anxiety Scale (HAMA). A lower score indicates less anxiety.
Change in Psychological Status (Depression) | Baseline, 12 weeks
  Assessed using the Hamilton Depression Scale (HAMD). A lower score indicates less depression.
Change in Quality of Life | Baseline, 12 weeks
  Measured using the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36), which assesses eight domains of health.
Change in Cardiac Index (CI) | Baseline, 12 weeks
  Assessed non-invasively to measure cardiac output relative to body surface area.
Adherence to Rehabilitation Program | Up to 12 weeks
  Calculated as the percentage of completed sessions out of the 36 total prescribed sessions for the HBTCR and CBCR groups.
Incidence of Major Adverse Events | Up to 12 weeks
  Number of participants experiencing major adverse cardiovascular events (e.g., death, myocardial infarction, urgent revascularization).
Change in Stroke Volume Index (SVI) | Baseline, 12 weeks
  Assessed non-invasively to measure the volume of blood pumped from the ventricle per beat relative to body surface area.
Change in Systemic Vascular Resistance Index (SVRI) | Baseline, 12 weeks
  Assessed non-invasively to measure the resistance to blood flow offered by all systemic vasculature, indexed to body surface area.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China